CLINICAL TRIAL: NCT00350922
Title: A Psychoeducation Trial for People With Chronic Stable Angina
Brief Title: A Clinical Trial of a Self-Management Education Program for People With Chronic Stable Angina
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Toronto (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 452639
Record Dates: First submitted 2006-07-08; First posted 2006-07-11 (Estimated); Last update posted 2006-07-11 (Estimated); Status verified 2005-11

CONDITIONS: Chronic Stable Angina
MeSH Terms: conditions — Angina, Stable

INTERVENTIONS:
Behavioral: Psychoeducation

SUMMARY:
The purpose of this clinical trial was to determine the effectiveness of a supportive and educational self-management program for improving health-related quality of life (HRQOL), angina symptoms, and self-efficacy and resourcefulness to self-manage for chronic angina patients. 130 participants were enrolled in the trial for 3 months. The program, entitled the Chronic Angina Self-Management Program, (CASMP) was found effective for improving HRQOL, angina symptoms, and self-efficacy to manage symptoms, compared to usual care.

ELIGIBILITY:
Inclusion Criteria:

Medical diagnosis of coronary artery disease CCS Class I-III Angina for at least 6 months Speak, read, understand English -

Exclusion Criteria:

MI/Bypass last 6 months CCS Class IV angina A major cognitive disorder -

Min Age: 0 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 130
Dates: Start 2003-09; Study Completion 2005-11

PRIMARY OUTCOMES:
SF36
Seattle Angina Questionnaire

SECONDARY OUTCOMES:
Self-Efficacy Scale
Self-Control Schedule

CONTACTS AND LOCATIONS:
Overall Officials: Judy H Watt-Watson, PhD, Study Director — University of Toronto; Michael H McGillion, PhD, Principal Investigator — University of Toronto
Locations (1):
- University of Toronto, Toronto, Ontario, Canada